CLINICAL TRIAL: NCT01067248
Title: Patho-physiology of Osteoporosis in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) and Osteoporosis
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Maastricht University Medical Center (Other); Center for Integrated Rehabilitation and Organ Failure Horn (Other)
Responsible Party: Principal Investigator, Lisette Romme, MD, PhD, Catharina Ziekenhuis Eindhoven
Other Study IDs: M09-1971
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Osteoporosis
Keywords: COPD; Osteoporosis; Pathophysiology; Mechanism; Bone markers; Bone turnover; Protein turnover; Ageing; Endocrinology; Vitamin D
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Markers of ageing, such as telomere length and sirtuin 1.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD, osteoporosis: The subjects are divided into 6 groups of 20 subjects each, I: COPD patients with osteoporosis based on T-score and without vertebral fractures, II: COPD patients with osteoporosis based on T-score and vertebral fractures, III: COPD patients with vertebral fractures and without osteoporosis based on T-score, IV: COPD patients without osteoporosis based on T-score and without vertebral fractures, V: healthy controls with osteoporosis based on T-score and without vertebral fractures, VI: healthy controls without osteoporosis based on T-score and without vertebral fractures.

SUMMARY:
The main objective is to study important factors in the patho-physiology of osteoporosis in patients with COPD. Therefore, the investigators will study biological markers in plasma and urine and correlate them to markers of bone turnover and clinical data.

DETAILED DESCRIPTION:
Rationale:

Chronic obstructive pulmonary disease (COPD) is defined as a preventable and treatable disease with significant extrapulmonary effects. Osteoporosis is recognized as one of these extrapulmonary consequences. It results in increased risk of fracture and thereby an increased morbidity and mortality. Nowadays it is believed that the patho-physiology of osteoporosis is multi-factorial. However, which factors are most important in patients with COPD is still not clear.

Objective:

The main objective is to study important factors in the patho-physiology of osteoporosis in patients with COPD. Therefore, we will study biological markers in plasma and urine and correlate them to markers of bone turnover and clinical data.

Study design:

The present study will be an observational, cross-sectional study.

ELIGIBILITY:
Inclusion Criteria for the COPD patients:

* Aged 50 years or older;
* Women have to be postmenopausal (amenorrhea for 12 months or more)
* COPD Global initiative of Obstructive Lung Disease (GOLD) I, II, III and IV according to the American Thoracic Society (ATS) guidelines;
* ≥ 12 pack years;
* No respiratory tract infection or exacerbation of the disease for at least 4 weeks before the study;
* No use of oral corticosteroids for at least 4 weeks before the study;
* No use of anti-osteoporotic medication (calcium, vitamin D, biphosphonates) before inclusion;
* Capable to provide informed consent.

Exclusion Criteria for the COPD patients:

* Malignancy in the last 5 years;
* Lung fibrosis;
* Inflammatory bowel disease;
* Rheumatoid arthritis;
* Alcohol abuse;
* Bronchiectasia;
* Auto immune diseases;
* Hypothyroidism or hyperthyroidism based on blood sampling for thyroid hormone (TSH, fT4).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In total 120 patients will be included. All subjects will be included from the outdoor clinic of the department of Pulmonology of the Catharina Hospital Eindhoven or Diagnostic Centre Eindhoven (DCE). The subjects are divided into 6 groups of 20 subjects each, I: COPD patients with osteoporosis based on T-score and without vertebral fractures, II: COPD patients with osteoporosis based on T-score and vertebral fractures, III: COPD patients with vertebral fractures and without osteoporosis based on T-score, IV: COPD patients without osteoporosis based on T-score and without vertebral fractures, V: healthy controls with osteoporosis based on T-score and without vertebral fractures, VI: healthy controls without osteoporosis based on T-score and without vertebral fractures.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emiel Wouters, MD, PhD, prof, Principal Investigator — Maastricht University Medical Center